CLINICAL TRIAL: NCT01547156
Title: Mobile Sipoo a Randomized Controlled Trial
Brief Title: Mobile Sipoo - Telemonitoring With Combined With Active Assistance Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VTT Technical Research Centre of Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MobileSipoo
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus Type 2; Hypertension
Keywords: patient decision support; telemonitoring; self-management; remote patient monitoring; active assistance technology; selfcare
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): Control group received usual care
- Telemonitoring group (Experimental): Intervention patients were given a remote patient monitoring toolbox that included a mobile telephone, software application, and assessment devices for measuring and remote reporting of hypertension and diabetes -related health parameters at home. The monitored parameters were body weight, steps, blood pressure and blood glucose. Based on their self-monitored data, patients received feedback that was automatically generated, theory-based, health promotion rich information that aimed at strengthening their self-care practices.
  Interventions: Device: Intervention group

INTERVENTIONS:
Device: Intervention group
  Arms: Telemonitoring group

SUMMARY:
Mobile Sipoo is a randomized controlled trial aiming to improve selfcare and outcomes of diabetes and hypertensive patients by introducing a remote patient monitoring system supported with automatic patient decision support. The feedback system is coupled with back-office health coaching.

DETAILED DESCRIPTION:
Self-monitored data from blood pressure meters (SMBP), glucometers (SMBG), scales and pedometers are transferred by mobile phone terminals to a tethered personal health record (PHR) integrated with the provider EHR. The PHR application includes tools to display of self-monitoring data.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of diabetes or hypertension made at least 6 months prior to inclusion to study.
* For hypertensive patients: Blood pressure over 140/90 mmHg (systolic and diastolic separately) treated or untreated
* Diabetes patients: Glycohemoglobin A1c over 6.5% but lower that 11%
* use of diabetes medication

Exclusion Criteria:

* Patients who decline to participate
* Patients specifically excluded by the health centre physician
* Patients unable to co-operate, expected poor study compliance (IT illiterate) or reluctance to perform self monitoring
* Pregnancy
* Patients with a life expectance of less than one year
* Patients with major elective surgery planned within 6 months or patient has had major surgery within last 2 months.
* Patients with psychiatric disorders (depression), abuse of alcohol or narcotics complicating or disabling participation in the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-05; Primary Completion 2012-03 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | 9 months
Change in Hba1c(for diabetes patients) | 9 months

SECONDARY OUTCOMES:
Achieving the desired target range | 9 months
  Target range for blood pressure is <= 135/85 mmHg. Target range for glycohemoglobin is <= 6.5%.
Adverse effects | 9 months
  hypotension, RR < 120/80 mmHg
Hypoglycemia | 9 months
  p-glucose < 3.5 mmol/l
Change in body weight | 9 months
Change in BMI | 9 months
Change in medication | 9 months
Change in FÍNSIK scores | 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sipoo Health Care Centre, Sipoo, Finland

REFERENCES:
- See also: Related Info — http://www.vtt.fi/sites/care4me/index.jsp?lang=en